CLINICAL TRIAL: NCT06529744
Title: Improving Prognostic Confidence in Neurodegenerative Diseases Causing Dementia Using Peripheral Biomarkers and Integrative Modeling
Acronym: CRND TorCA
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Baycrest (Other); Centre for Addiction and Mental Health (Other); Toronto Dementia Research Alliance (TDRA) (Unknown); University of Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, Principal Investigator, University Health Network, Toronto
Other Study IDs: 24-5283
Record Dates: First submitted 2024-04-29; First posted 2024-07-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Dementia; Alzheimer Disease; Dementia With Lewy Bodies; Vascular Dementia; Frontotemporal Dementia; Mild Cognitive Impairment; Corticobasal Syndrome; Progressive Supranuclear Palsy; Parkinson Disease; Primary Progressive Aphasia
Keywords: alzheimer's disease; dementia; dementia with lewy bodies; vascular dementia; frontotemporal dementia; mild cognitive impairment; corticobasal syndrome; progressive supranuclear palsy; parkinson's disease; primary progressive aphasia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Lewy Body Disease; Dementia, Vascular; Frontotemporal Dementia; Cognitive Dysfunction; Corticobasal Degeneration; Supranuclear Palsy, Progressive; Parkinson Disease; Aphasia, Primary Progressive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood (including plasma, serum, RNA, and DNA), skin biopsy, and cerebrospinal fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop a model to predict disease progression in a large cohort of patients across a variety of neurodegenerative diseases, including Mild Cognitive Impairment (MCI) and dementia due to any neurodegenerative disease, including Alzheimer's Disease (AD), Lewy Body Disease (LBD), Vascular Disease (VaD) and Frontotemporal lobar degeneration (FTLD).

DETAILED DESCRIPTION:
The goal of this study is to create a model to predict disease progression in patients with mild cognitive impairments and forms of dementia. To accomplish this, the current study will evaluate different tests including: brain imaging (MRI), body fluid samples (blood and cerebrospinal fluid), skin biopsy, cognitive ability, and behavioural questionnaires. The study team hopes that this information can be used to guide diagnosis and better predict disease progression in patients with mild cognitive impairment and and early dementia.

ELIGIBILITY:
Inclusion Criteria:

* Possible or probable diagnosis of MCI or early dementia
* Age 30-95
* Study partner who has some weekly contact with patient. Some of the neuropsychological assessment require collateral from close contacts to assess cognition and functioning. Since neurodegenerative diseases can be associated with reduced cognition, including reduced awareness of one's own impairments, participants will be assessed for their capacity to consent at all study visits.
* Must, in the opinion of the site investigator, be able to complete most study procedures.

Exclusion Criteria:

* Participants who are not able to complete the majority of assessments in the opinion of the PI are excluded from the study. Exclusion criteria are evaluated at the site investigator's discretion; if the site investigator believes that the participant's symptoms are due to causes other than neurodegeneration, despite the presence of an exclusionary condition, the investigator may overrule the exclusion.

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with a mild cognitive impairment or early stage dementia that are between the ages of 30-95 can participate in the study as long as they have a study partner who can answer questionnaires at their 3 study visits and can complete a majority of assessments.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Cognitive phenotype | Baseline, 6-month follow-up, 1-year follow-up
  Change in Toronto Cognitive Assessment (TorCA) scores out of 330, where lower scores indicate increasing cognitive impairments, and individual domains.

SECONDARY OUTCOMES:
Assessment of DNA methylation (DNAm) from bloodwork | Baseline
  Biological age from DNA methylation (DNAm) collected via bloodwork compared to chronological age.
Neurodegenerative protein levels in biofluids and skin biopsy | Baseline, 6-month follow-up, 1-year follow-up
  Differences in protein levels between neurodegenerative diagnoses and predictive ability for change in TorCA
Structural and Functional Differences between neurodegenerative diseases via MRI of the brain | Baseline
  Brain volumes and white matter hyperintensity (WMH) load corresponding to Toronto Cognitive Assessment (TorCA) scores out of 330 where lower scores indicate increasing cognitive impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Tartaglia, M.D., Principal Investigator — Toronto Western Hospital, UHN; Tanz CRND
Locations (4):
- Canada (4):
  - Baycrest, North York, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers. Only anonymized responses to the cognitive assessment, clinical assessment, behavioural questionnaires and biofluid protein levels will be shared.

REFERENCES:
- [Background] Robinson JL, Lee EB, Xie SX, Rennert L, Suh E, Bredenberg C, Caswell C, Van Deerlin VM, Yan N, Yousef A, Hurtig HI, Siderowf A, Grossman M, McMillan CT, Miller B, Duda JE, Irwin DJ, Wolk D, Elman L, McCluskey L, Chen-Plotkin A, Weintraub D, Arnold SE, Brettschneider J, Lee VM, Trojanowski JQ. Neurodegenerative disease concomitant proteinopathies are prevalent, age-related and APOE4-associated. Brain. 2018 Jul 1;141(7):2181-2193. doi: 10.1093/brain/awy146. PMID 29878075
- [Background] Frost GR, Jonas LA, Li YM. Friend, Foe or Both? Immune Activity in Alzheimer's Disease. Front Aging Neurosci. 2019 Dec 10;11:337. doi: 10.3389/fnagi.2019.00337. eCollection 2019. PMID 31920620
- [Background] Bergsma T, Rogaeva E. DNA Methylation Clocks and Their Predictive Capacity for Aging Phenotypes and Healthspan. Neurosci Insights. 2020 Jul 21;15:2633105520942221. doi: 10.1177/2633105520942221. eCollection 2020. PMID 32743556
- [Background] Zhang M, Tartaglia MC, Moreno D, Sato C, McKeever P, Weichert A, Keith J, Robertson J, Zinman L, Rogaeva E. DNA methylation age-acceleration is associated with disease duration and age at onset in C9orf72 patients. Acta Neuropathol. 2017 Aug;134(2):271-279. doi: 10.1007/s00401-017-1713-y. Epub 2017 Apr 24. PMID 28439722
- [Background] Zhang M, McKeever PM, Xi Z, Moreno D, Sato C, Bergsma T, McGoldrick P, Keith J, Robertson J, Zinman L, Rogaeva E. DNA methylation age acceleration is associated with ALS age of onset and survival. Acta Neuropathol. 2020 May;139(5):943-946. doi: 10.1007/s00401-020-02131-z. Epub 2020 Mar 7. No abstract available. PMID 32146547
- [Background] Thijssen EH, La Joie R, Wolf A, Strom A, Wang P, Iaccarino L, Bourakova V, Cobigo Y, Heuer H, Spina S, VandeVrede L, Chai X, Proctor NK, Airey DC, Shcherbinin S, Duggan Evans C, Sims JR, Zetterberg H, Blennow K, Karydas AM, Teunissen CE, Kramer JH, Grinberg LT, Seeley WW, Rosen H, Boeve BF, Miller BL, Rabinovici GD, Dage JL, Rojas JC, Boxer AL; Advancing Research and Treatment for Frontotemporal Lobar Degeneration (ARTFL) investigators. Diagnostic value of plasma phosphorylated tau181 in Alzheimer's disease and frontotemporal lobar degeneration. Nat Med. 2020 Mar;26(3):387-397. doi: 10.1038/s41591-020-0762-2. Epub 2020 Mar 2. PMID 32123386
- [Background] Janelidze S, Berron D, Smith R, Strandberg O, Proctor NK, Dage JL, Stomrud E, Palmqvist S, Mattsson-Carlgren N, Hansson O. Associations of Plasma Phospho-Tau217 Levels With Tau Positron Emission Tomography in Early Alzheimer Disease. JAMA Neurol. 2021 Feb 1;78(2):149-156. doi: 10.1001/jamaneurol.2020.4201. PMID 33165506
- [Background] Ashton NJ, Pascoal TA, Karikari TK, Benedet AL, Lantero-Rodriguez J, Brinkmalm G, Snellman A, Scholl M, Troakes C, Hye A, Gauthier S, Vanmechelen E, Zetterberg H, Rosa-Neto P, Blennow K. Plasma p-tau231: a new biomarker for incipient Alzheimer's disease pathology. Acta Neuropathol. 2021 May;141(5):709-724. doi: 10.1007/s00401-021-02275-6. Epub 2021 Feb 14. PMID 33585983
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Feldman HH, Frisoni GB, Hampel H, Jagust WJ, Johnson KA, Knopman DS, Petersen RC, Scheltens P, Sperling RA, Dubois B. A/T/N: An unbiased descriptive classification scheme for Alzheimer disease biomarkers. Neurology. 2016 Aug 2;87(5):539-47. doi: 10.1212/WNL.0000000000002923. Epub 2016 Jul 1. PMID 27371494
- [Background] Amor S, Puentes F, Baker D, van der Valk P. Inflammation in neurodegenerative diseases. Immunology. 2010 Feb;129(2):154-69. doi: 10.1111/j.1365-2567.2009.03225.x. PMID 20561356
- [Background] Cuyvers E, Sleegers K. Genetic variations underlying Alzheimer's disease: evidence from genome-wide association studies and beyond. Lancet Neurol. 2016 Jul;15(8):857-868. doi: 10.1016/S1474-4422(16)00127-7. PMID 27302364
- [Background] Woollacott IOC, Nicholas JM, Heller C, Foiani MS, Moore KM, Russell LL, Paterson RW, Keshavan A, Schott JM, Warren JD, Heslegrave A, Zetterberg H, Rohrer JD. Cerebrospinal Fluid YKL-40 and Chitotriosidase Levels in Frontotemporal Dementia Vary by Clinical, Genetic and Pathological Subtype. Dement Geriatr Cogn Disord. 2020;49(1):56-76. doi: 10.1159/000506282. Epub 2020 Apr 28. PMID 32344399
- [Background] Sims R, Hill M, Williams J. The multiplex model of the genetics of Alzheimer's disease. Nat Neurosci. 2020 Mar;23(3):311-322. doi: 10.1038/s41593-020-0599-5. Epub 2020 Feb 28. PMID 32112059
- [Background] Leonenko G, Baker E, Stevenson-Hoare J, Sierksma A, Fiers M, Williams J, de Strooper B, Escott-Price V. Identifying individuals with high risk of Alzheimer's disease using polygenic risk scores. Nat Commun. 2021 Jul 23;12(1):4506. doi: 10.1038/s41467-021-24082-z. PMID 34301930
- [Background] Silbert LC, Dodge HH, Perkins LG, Sherbakov L, Lahna D, Erten-Lyons D, Woltjer R, Shinto L, Kaye JA. Trajectory of white matter hyperintensity burden preceding mild cognitive impairment. Neurology. 2012 Aug 21;79(8):741-7. doi: 10.1212/WNL.0b013e3182661f2b. Epub 2012 Jul 25. PMID 22843262
- [Background] Gouw AA, Seewann A, van der Flier WM, Barkhof F, Rozemuller AM, Scheltens P, Geurts JJ. Heterogeneity of small vessel disease: a systematic review of MRI and histopathology correlations. J Neurol Neurosurg Psychiatry. 2011 Feb;82(2):126-35. doi: 10.1136/jnnp.2009.204685. Epub 2010 Oct 9. PMID 20935330
- [Background] Shim YS, Yang DW, Roe CM, Coats MA, Benzinger TL, Xiong C, Galvin JE, Cairns NJ, Morris JC. Pathological correlates of white matter hyperintensities on magnetic resonance imaging. Dement Geriatr Cogn Disord. 2015;39(1-2):92-104. doi: 10.1159/000366411. Epub 2014 Nov 8. PMID 25401390
- [Background] Snyder HM, Corriveau RA, Craft S, Faber JE, Greenberg SM, Knopman D, Lamb BT, Montine TJ, Nedergaard M, Schaffer CB, Schneider JA, Wellington C, Wilcock DM, Zipfel GJ, Zlokovic B, Bain LJ, Bosetti F, Galis ZS, Koroshetz W, Carrillo MC. Vascular contributions to cognitive impairment and dementia including Alzheimer's disease. Alzheimers Dement. 2015 Jun;11(6):710-7. doi: 10.1016/j.jalz.2014.10.008. Epub 2014 Dec 12. PMID 25510382
- [Background] Alosco ML, Sugarman MA, Besser LM, Tripodis Y, Martin B, Palmisano JN, Kowall NW, Au R, Mez J, DeCarli C, Stein TD, McKee AC, Killiany RJ, Stern RA. A Clinicopathological Investigation of White Matter Hyperintensities and Alzheimer's Disease Neuropathology. J Alzheimers Dis. 2018;63(4):1347-1360. doi: 10.3233/JAD-180017. PMID 29843242
- [Background] Grimmer T, Faust M, Auer F, Alexopoulos P, Forstl H, Henriksen G, Perneczky R, Sorg C, Yousefi BH, Drzezga A, Kurz A. White matter hyperintensities predict amyloid increase in Alzheimer's disease. Neurobiol Aging. 2012 Dec;33(12):2766-73. doi: 10.1016/j.neurobiolaging.2012.01.016. Epub 2012 Mar 10. PMID 22410648
- [Background] Whitwell JL, Avula R, Senjem ML, Kantarci K, Weigand SD, Samikoglu A, Edmonson HA, Vemuri P, Knopman DS, Boeve BF, Petersen RC, Josephs KA, Jack CR Jr. Gray and white matter water diffusion in the syndromic variants of frontotemporal dementia. Neurology. 2010 Apr 20;74(16):1279-87. doi: 10.1212/WNL.0b013e3181d9edde. PMID 20404309
- [Background] Zhang Y, Schuff N, Du AT, Rosen HJ, Kramer JH, Gorno-Tempini ML, Miller BL, Weiner MW. White matter damage in frontotemporal dementia and Alzheimer's disease measured by diffusion MRI. Brain. 2009 Sep;132(Pt 9):2579-92. doi: 10.1093/brain/awp071. Epub 2009 May 12. PMID 19439421
- [Background] Freedman M, Leach L, Carmela Tartaglia M, Stokes KA, Goldberg Y, Spring R, Nourhaghighi N, Gee T, Strother SC, Alhaj MO, Borrie M, Darvesh S, Fernandez A, Fischer CE, Fogarty J, Greenberg BD, Gyenes M, Herrmann N, Keren R, Kirstein J, Kumar S, Lam B, Lena S, McAndrews MP, Naglie G, Partridge R, Rajji TK, Reichmann W, Uri Wolf M, Verhoeff NPLG, Waserman JL, Black SE, Tang-Wai DF. The Toronto Cognitive Assessment (TorCA): normative data and validation to detect amnestic mild cognitive impairment. Alzheimers Res Ther. 2018 Jul 18;10(1):65. doi: 10.1186/s13195-018-0382-y. PMID 30021658
- [Background] Prive F, Vilhjalmsson BJ, Aschard H, Blum MGB. Making the Most of Clumping and Thresholding for Polygenic Scores. Am J Hum Genet. 2019 Dec 5;105(6):1213-1221. doi: 10.1016/j.ajhg.2019.11.001. Epub 2019 Nov 21. PMID 31761295
- [Background] Zhang M, Ferrari R, Tartaglia MC, Keith J, Surace EI, Wolf U, Sato C, Grinberg M, Liang Y, Xi Z, Dupont K, McGoldrick P, Weichert A, McKeever PM, Schneider R, McCorkindale MD, Manzoni C, Rademakers R, Graff-Radford NR, Dickson DW, Parisi JE, Boeve BF, Petersen RC, Miller BL, Seeley WW, van Swieten JC, van Rooij J, Pijnenburg Y, van der Zee J, Van Broeckhoven C, Le Ber I, Van Deerlin V, Suh E, Rohrer JD, Mead S, Graff C, Oijerstedt L, Pickering-Brown S, Rollinson S, Rossi G, Tagliavini F, Brooks WS, Dobson-Stone C, Halliday GM, Hodges JR, Piguet O, Binetti G, Benussi L, Ghidoni R, Nacmias B, Sorbi S, Bruni AC, Galimberti D, Scarpini E, Rainero I, Rubino E, Clarimon J, Lleo A, Ruiz A, Hernandez I, Pastor P, Diez-Fairen M, Borroni B, Pasquier F, Deramecourt V, Lebouvier T, Perneczky R, Diehl-Schmid J, Grafman J, Huey ED, Mayeux R, Nalls MA, Hernandez D, Singleton A, Momeni P, Zeng Z, Hardy J, Robertson J, Zinman L, Rogaeva E; International FTD-Genomics Consortium (IFGC). A C6orf10/LOC101929163 locus is associated with age of onset in C9orf72 carriers. Brain. 2018 Oct 1;141(10):2895-2907. doi: 10.1093/brain/awy238. PMID 30252044
- [Background] Zhang M, Xi Z, Saez-Atienzar S, Chia R, Moreno D, Sato C, Montazer Haghighi M, Traynor BJ, Zinman L, Rogaeva E. Combined epigenetic/genetic study identified an ALS age of onset modifier. Acta Neuropathol Commun. 2021 Apr 23;9(1):75. doi: 10.1186/s40478-021-01183-w. PMID 33892821
- [Background] Visanji NP, Ghani M, Yu E, Kakhki EG, Sato C, Moreno D, Naranian T, Poon YY, Abdollahi M, Naghibzadeh M, Rajalingam R, Lozano AM, Kalia SK, Hodaie M, Cohn M, Statucka M, Boutet A, Elias GJB, Germann J, Munhoz R, Lang AE, Gan-Or Z, Rogaeva E, Fasano A. Axial Impairment Following Deep Brain Stimulation in Parkinson's Disease: A Surgicogenomic Approach. J Parkinsons Dis. 2022;12(1):117-128. doi: 10.3233/JPD-212730. PMID 34602499
- [Background] Fischl B, van der Kouwe A, Destrieux C, Halgren E, Segonne F, Salat DH, Busa E, Seidman LJ, Goldstein J, Kennedy D, Caviness V, Makris N, Rosen B, Dale AM. Automatically parcellating the human cerebral cortex. Cereb Cortex. 2004 Jan;14(1):11-22. doi: 10.1093/cercor/bhg087. PMID 14654453
- [Background] Dale AM, Fischl B, Sereno MI. Cortical surface-based analysis. I. Segmentation and surface reconstruction. Neuroimage. 1999 Feb;9(2):179-94. doi: 10.1006/nimg.1998.0395. PMID 9931268
- [Background] Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. Proc Natl Acad Sci U S A. 2000 Sep 26;97(20):11050-5. doi: 10.1073/pnas.200033797. PMID 10984517
- [Background] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200
- [Background] Schmidt P, Gaser C, Arsic M, Buck D, Forschler A, Berthele A, Hoshi M, Ilg R, Schmid VJ, Zimmer C, Hemmer B, Muhlau M. An automated tool for detection of FLAIR-hyperintense white-matter lesions in Multiple Sclerosis. Neuroimage. 2012 Feb 15;59(4):3774-83. doi: 10.1016/j.neuroimage.2011.11.032. Epub 2011 Nov 18. PMID 22119648